CLINICAL TRIAL: NCT07214090
Title: Pilot Single-center, Randomized, Controlled Study Evaluating the Therapeutic Effects of Passive Exposure Virtual Reality on Pain, Anxiety, Fatigue, and Well-being in Patients With Complex Palliative Care Needs.
Brief Title: Pilot Study Evaluating the Therapeutic Effects of Passive Exposure Virtual Reality on Pain, Anxiety, Fatigue, and Well-being in Patients With Complex Palliative Care Needs.
Acronym: EPURAVAS
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9787
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Palliative Care
Keywords: Palliative care; Virtual Reality Exposure Therapy; Virtual Reality; Pain modulation; Clinical Efficacy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- RVAT: The RVAT group serves as the control against which the experimental RVEP method is measured. Individuals in this group use a headset that is designed to be transparent or augmented, allowing them to remain aware of and oriented to their actual environment-the room they are in. While they may see some minimal virtual elements, there is no escape or full immersion into an alternative reality.
  Interventions: Behavioral: Transparent Augmented Reality with Real-World Video Feed Overlay (RVAT)
- RVEP: Individuals in this group use a VR headset that creates a full sensory immersion, meaning the real world is completely blocked out. The experience involves being transported into calming, computer-generated environments, such as tranquil nature scenes. The goal of this full immersion is to achieve a deep, passive distraction that effectively shifts attention away from symptoms like pain and anxiety.
  Interventions: Behavioral: Passive Multisensory Virtual Reality Immersion via Head-Mounted Display (RVEP)

INTERVENTIONS:
Behavioral: Transparent Augmented Reality with Real-World Video Feed Overlay (RVAT) — This intervention uses a transparent augmented virtual reality headset equipped with forward-facing cameras that capture the patient's real-world environment in real time. Transparent virtual and augmented reality overlays computer-generated elements (e.g., visual cues, guidance, or interactive content) onto the live view of the physical environment. This approach maintains a strong anchoring in reality while providing therapeutic visual enhancements, tailored in real-time to the patient's responses. Sessions last 10 minutes and are delivered in a controlled clinical environment, supervised by trained staff.
  Groups: RVAT
Behavioral: Passive Multisensory Virtual Reality Immersion via Head-Mounted Display (RVEP) — This intervention involves the use of a head-mounted display to immerse the patient in a fully computer-generated virtual environment. The virtual reality passive exposure is designed to distract patients from painful or anxiety-inducing sensations by engaging multiple sensory modalities (visual, auditory, and occasionally tactile). Patients are exposed to relaxing or engaging scenarios, such as natural landscapes or calm immersive scenes, without requiring interaction. Sessions last 10 minutes and are delivered in a controlled clinical environment, supervised by trained staff.
  Groups: RVEP

SUMMARY:
The EPURAVAS "Pilot Study Using Augmented and Virtual Reality to Ease Suffering in Palliative Care" study is designed to investigate a non-medication treatment for complex symptoms in palliative care.

The purpose is to assess the clinical effectiveness of Virtual Reality (VR) exposure as a way to relieve the distressing symptoms experienced by individuals receiving specialized palliative care.

The study seeks to determine if immersive Passive Exposure Virtual Reality (RVEP) is more effective at providing a significant reduction in pain and anxiety, and a greater overall improvement in well-being and quality of life for patients in complex palliative situations, compared to a control virtual reality approach.

In the study, individuals are randomly assigned to one of two groups for a week:

* Immersive VR: A headset completely surrounds the user in a calming, computer-generated world, aiming to deeply distract the mind from discomfort.
* Control VR: A different headset allows the user to still see the real room while potentially having some virtual elements added. This acts as a comparison to measure the specific benefits of the deep immersion.

Participation involves daily 10-minute VR sessions for seven days. Throughout this time, physiological measurements are safely and continuously recorded using the VR headset and a connected watch. This collects objective information on how the body is reacting-things like brain activity, heart rate, and breathing-to scientifically determine the treatment's impact.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Hospitalized in the palliative care unit or followed by the mobile palliative care team of the Strasbourg University Hospitals
* Estimated life expectancy > 1 month (Pronopall score calculated based on medical record data)
* Affiliated with a social security scheme
* Able to understand the objectives and risks of the trial
* Able to understand and complete study questionnaires written in French
* Reachable by phone or email for the entire duration of participation in the study

Exclusion Criteria:

* Patient with a psychotic mental illness, followed and treated before the study, and not stabilized
* Patient with a severe neurological disease, followed and treated before the study, and not stabilized
* Patient with visual or auditory disorders, or motion sickness, present before the study, that could interfere with the use of virtual reality
* Patient under legal protection or unable to express their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from the palliative care unit or through the mobile palliative care team at Strasbourg University Hospitals.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Effectiveness Assessed by ESAS F12 Pain Score | Day 0 (J0) to Day 7 (J7)
  Clinical effectiveness of the RVEP and RVAT interventions will be evaluated using the ESAS F12 questionnaire. A clinically significant improvement is defined as a reduction of at least 2 points on the numeric pain scale between Day 0 and Day 7. Each subject will be classified as "effective" (yes/no) based on this criterion, allowing comparison of effectiveness percentages between groups.

SECONDARY OUTCOMES:
Presence of Pain Assessed by EEG | During each session from Day 0 to Day 7
  Pain presence will be evaluated using EEG recordings during each session. A pain episode is defined as Piq ≥10%. This outcome assesses the physiological signal of pain during RVEP and RVAT sessions.
Pain Experience Assessed by the French Short Version of the Brief Pain Inventory (QCD in french, or BPI in english) | Before the first session, Day 7 (J7), and Day 14 (J14)
  Pain experience will be tracked using the BPI questionnaire to evaluate changes in the subjective experience of pain from baseline through Day 14.
  Certainly, here is a brief description of the three assessment scales you've asked about:
  The BPI is a comprehensive, self-report tool designed to assess both the intensity of a patient's pain and the degree to which that pain interferes with their daily life. The patient uses a 0 to 10 scale to rate pain severity (e.g., worst, least, and average pain) and the impact on seven different activities (like mood, walking, and sleep). The BPI is typically analyzed as two separate average scores-Pain Severity and Pain Interference-to provide a clear picture of the pain's physical and functional dimensions. Higher scores indicate a worse outcome, meaning more intense pain or greater functional interference.
Dropout and Exclusion Rate | Day 0 to Day 14
  The percentage of participants lost to follow-up or excluded during the study will be calculated in order to assess protocol feasibility and support future sample size calculations for comparative studies.
Emotional and Functional Outcomes - Objective Physiological Data | Continuously during each session from Day 0 to Day 7
  Physiological data will be collected from EEG (electroencephalography) via KAPTICS© headset, and Embrace Plus© smartwatches to assess functional and emotional responses to RV interventions.
  EEG measures the electrical activity of the brain. The raw data is recorded as voltage fluctuations over time.
Discomfort Symptoms Assessed by ESAS F12 | Before and after each session from Day 0 to Day 7
  The ESAS F12 ( Edmonton Symptom Assessment System) questionnaire will be used to assess self-reported symptoms of discomfort before and after each session.
  Minimum Value: The minimum possible score is 0. Maximum Value: The maximum possible score is 120. Interpretation of Scores: Higher scores mean a worse outcome or greater severity of the symptom. A score of 0 means the symptom is absent ("no pain," "not tired"), and a score of 120 means the symptom is at its "worst possible severity."
Anxiety Symptoms Assessed by HADS-A | Before and after each session until Day 7, and again at Day 14
  Anxiety levels will be measured using the anxiety subscore ("A") of the Hospital Anxiety and Depression Scale (HADS) to evaluate changes in emotional state throughout the intervention period.
  Scores on the HADS scale (Hospital Anxiety and Depression Scale) for anxiety symptoms. Structure: 14 items total, split into two subscales: - HADS-A (Anxiety) - 7 items - HADS-D (Depression) - 7 items Minimum value: 0 (no symptoms). Maximum value: 21 per subscale (if all items scored at the maximum of 3). but 42 total if both subscales are summed. Interpretation: Higher scores reflect a worse outcome, meaning greater anxiety and/or depressive symptom severity.
Well-Being Assessed by WHO-5 Well-Being Index (OMS-5 in french) | Day 0 (J0), Day 7 (J7), and Day 14 (J14)
  Subjective well-being will be assessed using the WHO-5 questionnaire to track changes in psychological health over time.
  The WHO-5 Well-Being Index is a short, simple questionnaire that measures a person's current mental well-being and is primarily used to screen for depression.
  This scale consists of just five questions that ask the patient to rate how often they have felt a certain way over the past two weeks (e.g., cheerful, calm, full of energy). Each item is scored on a scale from 0 (at no time) to 5 (all the time). The total raw score is calculated by summing the five item scores, which is then multiplied by four to create a final score between 0 and 100.
Fatigue Assessed by the Multidimensional Fatigue Inventory (MFI-20) | Day 0 (J0), Day 7 (J7), and Day 14 (J14)
  The MFI-20 questionnaire will evaluate multidimensional fatigue to assess physical and mental fatigue trajectories throughout the study.
  The MFI-20 questionnaire is the Multidimensional Fatigue Inventory. Minimum Value (per subscale): 4 Maximum Value (per subscale): 20 The MFI-20 is composed of five subscales (General Fatigue, Physical Fatigue, Reduced Activity, Reduced Motivation, and Mental Fatigue), each with a score range of 4 to 20. The use of a single total score over all 20 items is generally not recommended. Higher scores on the MFI-20 reflect more severe or greater fatigue, meaning a worse outcome.
Tolerance of VR Exposure - Cybersickness Symptoms | Before and after each session from Day 0 to Day 7
  Cybersickness symptoms will be monitored using the VRISE-fr scale to evaluate tolerance to virtual reality exposure during the intervention.
  The "VRISE-fr" scale stands for Virtual Reality-Induced Symptoms and Effects (French adaptation).
  Minimum Value: 0 (No symptoms). Maximum Value: 35 Interpretation: Higher scores mean a worse outcome (greater severity of symptoms/sickness).
Subjective Experience of Intervention - Semi-Structured Interview | Day 14 (J14)
  A semi-structured interview will be conducted using a guide with five open-ended questions to qualitatively assess the participant's experience and perception of the intervention.
Emotional and Functional Outcomes - Objective Physiological Data | Continuously during each session from Day 0 to Day 7
  Physiological data will be collected from EOG (electrooculography) via KAPTICS© headset, and Embrace Plus© smartwatches to assess functional and emotional responses to RV interventions.
  The EOG data is primarily used to track and quantify eye movements

IPD SHARING:
Plan to Share IPD: Undecided